CLINICAL TRIAL: NCT02372136
Title: Individualizing and Optimizing Nutrition to Prevent Metabolic Syndrome and To Improve Neurodevelopment in Preterm and Small for Gestational Age Infants
Brief Title: Optimizing Individual Nutrition in Preterm Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other); The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Luc P. Brion, MD, Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 102014-056
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Infant, Premature, Diseases; Infant, Small for Gestational Age
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the statistician and the formula technicians know the patients' allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized and Optimized Nutrition (Experimental): Individualized nutrition Optimized nutrition
  Interventions: Dietary Supplement: Individualized Nutrition; Dietary Supplement: Optimized nutrition
- Optimized Nutrition (Other): Optimized nutrition
  Interventions: Dietary Supplement: Optimized nutrition

INTERVENTIONS:
Dietary Supplement: Individualized Nutrition — Intake of macronutrients (protein, fat, and carbohydrate) will be individualized every day by adding one or more macronutrients to human milk based on daily measurements using near-infrared analysis.
  In patients receiving less milk than 140 ml x kg-1 x day-1 fortification of human milk will be adjusted to reach at least the average concentrations of protein, fat, and carbohydrate in donor's milk (Wojcik. J Am Diet Assoc. 2009 Jan;109:137-40) and 20 cal/oz as provided by the Mother's Milk Bank of North Texas.
  In those receiving at least 140 ml x kg-1 x day-1 of milk at 24 cal/oz fortification will be adjusted to meet recent guidelines from the the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition (ESPGHAN) (Agostoni et al. J Pediatr Gastroenterol Nutr. 2010 Jan;50:85-91).
  Other Names: Targeted, customized
  Arms: Individualized and Optimized Nutrition
Dietary Supplement: Optimized nutrition — Milk fortification will be based on current recommendations and optimized by adjustment of nutrients once a week based on blood levels of urea nitrogen (corrected for serum creatinine level) and albumin and velocity of growth (weight and length).
  Other Names: Adjustable

SUMMARY:
In preterm infants fed human milk, milk needs to be fortified to meet nutrient recommendations. Fortification can be 1) standard, 2) individualized (adjusted based on daily human milk nutrient analysis and milk volume), or 3) optimized (adjusted based on growth rate and serum analyses).

The first specific aim will determine whether individualized and optimized nutrition during hospitalization results in improved growth in the neonatal intensive care unit (NICU) in extremely low gestational age (GA) neonates (ELGANs, <29 weeks) and in small for GA (SGA, birth weight <10th percentile for GA) preterm infants compared with optimized nutrition.

The second specific aim will determine whether individualized and optimized nutrition in the NICU improves neurodevelopmental outcomes (acquisition of development milestones) and reduces the risk of disproportionate growth (i.e., excess fat) in the NICU and findings suggestive of metabolic syndrome in the first 3 years of life.

DETAILED DESCRIPTION:
Hypotheses:

1. Primary hypothesis: In preterm infants (GA <29 weeks or GA <35 weeks and SGA) individualized and optimized nutrition will increase velocity of growth (weight gain velocity by 2 g x kg-1 x day-1 and length velocity by 0.2 cm per week) from birth to 36 weeks of postmenstrual age (GA plus postnatal age) or discharge (whichever comes first) in comparison with optimized nutrition.
2. Secondary hypotheses: Individualized and optimized nutrition will improve neurodevelopmental outcome and reduce the risk of disproportionate growth (excess fat) in the NICU and findings suggestive of metabolic syndrome in the first 3 years of life.

Study design:

Double-blinded randomized controlled trial (RCT): After consent, 150 neonates will be randomized to one of two groups.

Study intervention: Patients will be randomized to either:

1. Control: optimized nutrition: Milk fortification will be based on current recommendations and optimized by adjustment of nutrients once a week based on blood levels of urea nitrogen and albumin and velocity of growth (weight and length).
2. Intervention: Individualized and optimized nutrition: Milk fortification will be optimized as in control neonates. In addition, nutrition will be individualized every day. Milk fortification will be adjusted based on daily measurements of macronutrients in human milk using near-infrared analysis.

Randomization will be done by computer provided by a statistician using random block allocation and stratification by GA and size for age (AGA [appropriate for GA] 23-28 weeks, SGA 23-28 weeks and SGA 29-34 weeks). Twins and multiples will be randomized to the same arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <29 weeks GA and SGA infants <35 weeks GA born at Parkland Health and Hospital System
* Maternal plan to breastfeed or to use milk from the donor milk bank
* From birth to 1 week of life

Exclusion Criteria:

* Patients on comfort care only
* Patients with major congenital abnormalities
* Patients who are too unstable for the first 7 days to have an accurate length measurement

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc P Brion, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study will be available from the corresponding author on reasonable request after completion and publication of all follow-up data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after completion and publication of all follow-up data
Access Criteria: on reasonable request

REFERENCES:
- [Background] Brion LP, Rosenfeld CR, Heyne R, Brown LS, Lair CS, Petrosyan E, Jacob T, Caraig M, Burchfield PJ. Optimizing individual nutrition in preterm very low birth weight infants: double-blinded randomized controlled trial. J Perinatol. 2020 Apr;40(4):655-665. doi: 10.1038/s41372-020-0609-1. Epub 2020 Feb 18. PMID 32071367
- [Derived] Reis JD, Heyne R, Rosenfeld CR, Caraig M, Brown LS, Burchfield PJ, Lair CS, Petrosyan E, Jabob T, Nelson DB, Brion LP. Follow-up of a randomized trial optimizing neonatal nutrition in preterm very low birthweight infants: growth, serum adipokines, renal function and blood pressure. J Perinatol. 2024 Jan;44(1):78-86. doi: 10.1038/s41372-023-01821-2. Epub 2023 Nov 14. PMID 37964083
- [Derived] Reis JD, Tolentino-Plata K, Caraig M, Heyne R, Rosenfeld CR, Brown LS, Brion LP. Double-blinded randomized controlled trial of optimizing nutrition in preterm very low birth weight infants: Bayley scores at 18-38 months of age. J Perinatol. 2023 Jan;43(1):81-85. doi: 10.1038/s41372-022-01572-6. Epub 2022 Dec 6. PMID 36473929
- See also: DOI — https://DOI.org/10.1038/s41372-020-0609-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Preterm neonates born at Parkland Hospital between January 27, 2016 and September 10, 2018
Pre-assignment Details: Neonates were excluded if they received comfort care only, had a major congenital abnormality, or were too unstable for the ﬁrst 7 days to have an accurate length measurement using a length board or a caliper.
Groups:
- Individualized and Optimized Nutrition: Individualized nutrition Optimized nutrition
  Individualized Nutrition: Intake of macronutrients (protein, fat, and carbohydrate) will be individualized every day by adding one or more macronutrients to human milk based on daily measurements using near-infrared analysis.
  In patients receiving less milk than 140 ml x kg-1 x day-1 fortification of human milk will be adjusted to reach at least the average concentrations of protein, fat, and carbohydrate in donor's milk (Wojcik. J Am Diet Assoc. 2009 Jan;109:137-40) and 20 cal/oz as provided by the Mother's Milk Bank of North Texas.
  In those receiving at least 140 ml x kg-1 x day-1 of milk at 24 cal/oz fortification will be adjusted to meet recent guidelines from the the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition (ESPGHAN) (Agostoni et al. J Pediatr Gastroenterol Nutr. 2010 Jan;50:85-91).
  Optimized nutrition: Milk fortification will be based on current recommendations and optimized by adjustment of nutrients once a week based on blood levels of urea nitrogen (corrected for serum creatinine level) and albumin and velocity of growth (weight and length).
Period: Overall Study
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Started | 62 | 58
Completed | 59 | 57
Not Completed | 3 | 1
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Individualized and Optimized Nutrition: Both individualized and optimized nutrition
- Optimized Nutrition: Optimized nutrition only
- Total: Total of all reporting groups
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 28 (3) | 28 (3) | 28 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 31 | 25 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 39 | 80
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 45 | 40 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Birth weight [Mean (Standard Deviation); unit: grams] | 1024 (304) | 1034 (294) | 1029 (299)
Birth length [Mean (Standard Deviation); unit: cm] — Population: Accurate validated birth length was not obtained in 4 newborns.
  cm
    number analyzed (Participants) | 59 | 57 | 116
    (all) | 35.6 (3.6) | 35.5 (3.4) | 35.6 (3.5)
Birth fronto-occipital circumference [Mean (Standard Deviation); unit: cm] | 24.7 (2.4) | 24.9 (2.5) | 24.8 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Growth Velocity
Description: Rate of weight gain [g x kg-1 x day-1] and length velocity [cm x week-1]
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Measure: Mean (Standard Deviation); unit: g kg-1 day-1
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 59 | 57
g kg-1 day-1 | 13 (2.6) | 13.1 (2.1)

2. Primary Outcome: Linear Growth Velocity
Description: Increase in body length per week from birth to 36 weeks postmenstrual age or discharge
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Data were not available for patients transferred to another institution
Measure: Mean (Standard Deviation); unit: cm per week
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 52 | 55
cm per week | 0.90 (0.23) | 0.91 (0.18)

3. Secondary Outcome: Disproportionate Growth (Increased Fat Mass): BMI >90th Centile
Description: Disproportionate growth (increased fat mass): BMI > 90th centile for sex and age
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Total number is limited by need for accurate validated length and weight on the same day. This was not available in patients who were transferred.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 50 | 55
Participants | 1 | 1

4. Secondary Outcome: Blood Pressure
Description: Systolic blood pressure (calm or sleeping)
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 50 | 50
mm Hg | 69.4 (7.2) | 69.7 (6.9)

5. Secondary Outcome: Hypertension or High Systolic Blood Pressure
Description: Systolic blood pressure >90th centile defined by the SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN
Time Frame: at 33-48 months adjusted age
Population: 33-48 months adjusted age Not all participants entered follow-up and had data collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 40 | 38
Participants | 7 | 3

6. Secondary Outcome: Neurodevelopment
Description: Bayley Scale of Infant and Toddler Development, Third Edition (BSID-III): cognitive composite score Higher scores mean a better outcome. The composite scaled score has a mean of 100 and a SD of 15, a floor of 55 and a ceiling of 145.
  Bayley, N. (2006). Bayley Scales of Infant and Toddler Development- Third Edition. San Antonio, TX: Harcourt Assessment.
  DOI: 10.1177/0734282906297199
Time Frame: 18-41 months adjusted age (postnatal age corrected for prematurity)
Population: BSID-III assessment was performed at 18-38 months of age corrected for prematurity, scored for corrected age, and adjusted for age of administration
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 47 | 44
score on a scale | 85 [75 to 90] | 85 [75 to 90]

7. Secondary Outcome: Neurodevelopment
Description: Bayley Scale of Infant and Toddler Development, Third Edition (BSID-III): language composite score Higher scores mean a better outcome. The composite scaled score has a mean of 100 and a SD of 15, a floor of 47 and a ceiling of 153.
  Bayley, N. (2006). Bayley Scales of Infant and Toddler Development- Third Edition. San Antonio, TX: Harcourt Assessment.
  DOI: 10.1177/0734282906297199
Time Frame: 18-41 months adjusted age (postnatal age corrected for prematurity) 18-41 months adjusted age (postnatal age corrected for prematurity) 18-41 months corrected age 18-41 months
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 47 | 44
score on a scale | 74 [68 to 84] | 74 [68 to 89]

8. Secondary Outcome: Leptin
Description: Serum levels of leptin (measure of adiposity)
Time Frame: 33-48 months adjusted age
Population: 33-48 months adjusted age Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 33 | 28
ng/ml | 2.8 (0.48) | 1.9 (0.32)

9. Secondary Outcome: Renal Function
Description: Serum level of cystatin C. This value increases if renal glomerular filtration decreases.
Time Frame: 33-48 months adjusted age
Population: 33-48 months adjusted age Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 36 | 32
mg/dl | .79 (.14) | .83 (.14)

10. Secondary Outcome: Comparison of Weight With Expected Value for Age and Gender
Description: Comparison of weight with expected value for age and gender: Z score for weight Expected mean for age and gender is zero. Normal is -2 to +2. Best is zero with concomitant zero for length.
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 59 | 57
Z-score | -1.05 (.9) | -1.18 (.8)

11. Secondary Outcome: Comparison of Length With Expected Value for Age and Gender
Description: Comparison of length with expected value for age and gender: Z score for length Expected mean for age and gender is zero. Normal is -2 to +2. Best is zero with concomitant zero for weight.
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 52 | 55
Z-score | -1.48 (0.9) | -1.61 (.9)

12. Secondary Outcome: Comparison of Head Size With Expected Value for Age and Gender
Description: Comparison of head size with expected value for age and gender: Z score for fronto-occipital circumference Expected mean for age and gender is zero. Normal is -2 to +2. Best is zero.
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 58 | 57
Z-score | -1.06 (1) | -1.24 (.9)

13. Secondary Outcome: Rate of Weight Gain
Description: Rate of weight gain
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 59 | 57
g/kg/day | 13 (2.6) | 13.1 (2.1)

14. Secondary Outcome: Rate of Linear Growth
Description: Rate of linear growth
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 52 | 55
cm/week | .9 (.23) | .91 (.18)

15. Secondary Outcome: Comparison of Rate of Head Growth With Expected Value for Age and Gender
Description: Change in z score for fronto-occipital circumference from birth to endpoint Expected mean for age and gender is zero. Normal is -2 to +2.
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Not all participants entered follow-up and had data collected.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 58 | 57
Z-score | -.63 (1) | -.74 (1.1)

16. Secondary Outcome: Body Composition
Description: Percent fat mass measured by Dexascan
Time Frame: at 1 year of age and 3 years of age
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Mortality
Description: Percent of infants who died from birth to endpoint (36 weeks post menstrual age or discharge from the neonatal intensive care unit if earlier than 36 weeks)
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 62 | 58
Participants | 3 | 1

18. Other Pre Specified Outcome: Necrotizing Enterocolitis
Description: Percentage of infants who developed necrotizing enterocolitis stage II or greater (using the modified Bell stage classification) in the neonatal intensive care unit
Time Frame: 36 (range 35-37) weeks postmenstrual age or discharge (whichever comes first)
Population: Until 36 weeks postmenstrual age or discharge from the neonatal intensive care unit if earlier than 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized and Optimized Nutrition | Optimized Nutrition
Number analyzed (Participants) | 62 | 58
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: from birth to discharge from the neonatal intensive care unit
Groups:
- Experimental: Optimized and individualized nutrition
- Control: Optimized nutrition
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 3/62 | 4/58
Serious Adverse Events (participants affected / at risk) | 6/62 | 5/58
Other Adverse Events (participants affected / at risk) | 19/62 | 17/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=62) | Control (N=58)
Necrotizing enterocolitis (Gastrointestinal disorders) | 6 (62) | 5 (58) — Necrotizing enterocolitis stage II or greater (modified Bell's classification)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=62) | Control (N=58)
Feeding intolerance (Gastrointestinal disorders) | 19 (62) | 17 (58) — Feeding intolerance (feeds held for 24 h for abdominal distention, vomiting or residuals)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02372136/Prot_SAP_000.pdf